CLINICAL TRIAL: NCT05858983
Title: A Multi-center, Open-label, Dose-escalation Phase I/II Clinical Study to Evaluate the Safety, Tolerability and Efficacy of FT-001 Administered Via Subretinal Injection in Subjects With Biallelic RPE65 Mutation-associated Retinal Dystrophy
Brief Title: Gene Therapy in Subjects With Biallelic RPE65 Mutation-associated Retinal Dystrophy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT001-C101
Record Dates: First submitted 2023-04-29; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-10

CONDITIONS: Biallelic RPE65 Mutation-associated Retinal Dystrophy
Keywords: FT-001; Biallelic RPE65 Mutation-associated Retinal Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FT-001 Dose 1 (Experimental): Intraocular administration of a single low dose of range FT-001
  Interventions: Genetic: FT-001 Low Dose
- FT-001 Dose 2 (Experimental): Intraocular administration of a single Mid dose of range FT-001
  Interventions: Genetic: FT-001 Mid Dose
- FT-001 Dose 3 (Experimental): Intraocular administration of a single High dose of range FT-001
  Interventions: Genetic: FT-001 High Dose

INTERVENTIONS:
Genetic: FT-001 Low Dose — Comparison of different dosages of FT-001
  Arms: FT-001 Dose 1
Genetic: FT-001 Mid Dose — Comparison of different dosages of FT-001
  Arms: FT-001 Dose 2
Genetic: FT-001 High Dose — Comparison of different dosages of FT-001
  Arms: FT-001 Dose 3

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and efficacy of subretinal administration of FT-001 in subjects with biallelic RPE65 mutation-associated retinal dystrophy.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, phase I/II clinical study to evaluate the safety, tolerability, efficacy, immunogenicity, and in vivo biodistribution characteristics of FT-001 in subjects with biallelic RPE65 mutation-associated retinal dystrophy. Assessments will include visual acuity, vector shedding, immunogenicity and adverse events. Participants will be monitored for 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and sign the ICF
2. Female or male aged 8-45 years old when signing the ICF
3. Clinically diagnosed with biallelic RPE65 mutation-associated retinal dystrophy

Exclusion Criteria:

1. Other interfering eye diseases
2. Presence of any systemic or ocular disease that can cause or likely to cause vision loss
3. There is evidence of obviously uncontrolled concomitant diseases
4. Known to have active or suspected autoimmune diseases
5. With active systemic infection under treatment
6. Pregnant or lactating women
7. Other conditions unsuitable for the study as determined by the investigator

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of FT-001(incidence of ocular and non-ocular AEs and SAEs) | 52 weeks
  Incidence of ocular and non-ocular AEs and SAEs

SECONDARY OUTCOMES:
Changes in visual function from baseline | 52 weeks
  Changes in visual function from baseline as assessed by FST
Changes in visual function from baseline | 52 weeks
  Changes in visual function from baseline as assessed by Mobility courses

CONTACTS AND LOCATIONS:
Overall Officials: Ruifang Sui, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No